CLINICAL TRIAL: NCT04822753
Title: A Randomized Placebo-Controlled Trial of Platelet Rich Plasma (PRP) for Facet Mediated Lumbar Low Back Pain
Brief Title: Platelet Rich Plasma (PRP) for Facet Mediated Lumbar Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WAMC.2021.0053
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Facet Joint Pain; Low Back Pain
Keywords: platelet rich plasma (PRP); Facet Joint; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded, assessor blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma injection to lumbar facet joint (Experimental): Platelet Rich Plasma injection to lumbar facet joint
  Interventions: Procedure: Platelet Rich Plasma injection to the lumbar facet joint
- Placebo injection to lumbar facet joint (Placebo Comparator): Placebo injection to lumbar facet joint
  Interventions: Procedure: Platelet Rich Plasma injection to the lumbar facet joint

INTERVENTIONS:
Procedure: Platelet Rich Plasma injection to the lumbar facet joint — Using standard fluoroscopic view, place a needle at the target facet joint. Inject about 1ml of study injectate.

SUMMARY:
Low back pain (LBP) is both the single most common cause of disability and the leading cause of visits when military personnel go to their primary care doctors. Military personnel that deal with LBP can often be placed on limited duty profile. Not surprisingly, the direct and indirect costs of low back and neck pain accounts for approximately $88 billion of health care expenditure. In order to reduce the large financial and personal cost, clinical studies must be designed to treat LBP. This study will provide evidence-based medicine on a new regenerative medicine treatment option that may significantly affect military personnel with LBP. PRP (Platelet Rich Plasma) may offer alternate treatment methods that may help preserve the facet joint structures, and improve pain and function without causing destructive lesions or worsening degenerative joints. This healing process may favor improved participation with rehabilitation therapy and ultimately improve return to duty status. This study will also assess the effectiveness of point of care generated PRP, as a minimally invasive treatment option for treating lumbar facet pain. Specifically, PRP effectiveness will be compared to injecting placebo control when injected into facet joints.

DETAILED DESCRIPTION:
This randomized controlled trial will determine the efficacy of platelet rich plasma vs. Control/Placebo. 170 healthy, physically active individuals with facet mediated lumbar low back pain will be recruited to participate in the study. Part of the formal screening procedures, consented participants will undergo a fluoroscopic guided diagnostic lumbar medial branch block (MBB) within 60 days after consent. The results of the diagnostic MBB will determine if they meet final eligibility criteria (facetogenic pathology) and should continue on with the therapeutic injection. In the rare case that there is a positive MBB within the past three months, then it will not be repeated. To clarify, the diagnostic MBB will determine if the procedure will be beneficial to the participant by confirming they have facet-mediated low back pain and that the experimental procedure may benefit them. This avoids participants continuing in the study who would not benefit from the PRP injection.

Participants will be asked to complete a standard pain diary following the lumbar MBB procedure. Participants who experience a positive test result from the MBB (as indicated by a reduction of ≥50% in pain symptoms using the 8 hour pain diary) will be eligible to proceed with the study. Following the stated inclusion/exclusion criteria, participants who do not experience a positive test result (indicate a reduction < 50% in pain symptoms) will be formally withdrawn from the study at this point and will resume normal care with their referring physician to explore their best treatment option(s).

Any female participant of child-bearing age will also be required to have a urine hCG test performed prior to the diagnostic or therapeutic injection being performed. If the urine hCG indicates the participant is pregnant, per stated inclusion/exclusion criteria, they will be formally withdrawn from the study at this point and will resume normal care with their referring provider.

Participants who meet final eligibility criteria (positive lumbar MBB and, if applicable, negative pregnancy test) will be randomized to a study arm within one week of the MBB. A computer-generated randomization program prepared by the study biostatistician will be used to assign participants 1:1 across both study arms (PRP vs. Control/Placebo).

The target area for either the PRP or saline injection will be the intra-articular facet joint. During this time, adequate amount of peripheral blood will be drawn by a clinic nurse; either 30ml if injecting single side, or 60ml will be drawn if injecting both sides. PRP mixture will be prepared using a point of care centrifuge system. Participants in the PRP group will receive 1 ml of PRP mixture for each facet joint. Participants in the control/placebo group will receive 1 ml of normal saline for each facet joint.

In order to facilitate blinding, both groups will have at least 30ml of blood drawn on the same day as the injection (PRP or saline). The blood drawn from participants in the control group will be safely discarded per standard protocols. For the PRP group, a small sample will be processed by point of care cell counter located within the Pain Clinic to establish baseline platelet, white blood cell, and hemoglobin level and hematocrit of the peripheral blood. In addition, a small sample of the actual prepared PRP solution will be processed to check for concentrated platelet, white blood cell and hemoglobin level.

All participants will be instructed to avoid other invasive treatments (including acupuncture) while participating in this study. In order to prevent a potential blunting-effect of the PRP treatment, participants will also be instructed to avoid non-emergent use of NSAIDs for treating typical pain symptoms for at least the first 3-months following the study intervention/injection to help the patient accurately reflect their perception of pain. NSAIDs may reduce the effectiveness of PRP. If a participant needs additional analgesia, acetaminophen is the preferred agent. Concomitant medications will be recorded at each follow up visit. If necessary, participants will received pain medication that is provided as SOC post-procedure.

Patients will be given appropriate temporary profile (if active duty) to protect them from aggravating activities (such as airborne operation, ruck marches, formation running for at least 3 months after the injection. All patients will be ask to enroll in pre and post procedure physical therapy sessions for body mechanics training/rehabilitative protocol, for total of up to 8 sessions during the study period. Participants will be evaluated by experienced physical therapist specializing in chronic pain. The pre-procedure rehabilitation will occur within a week prior to the procedure. The 1st post-procedure rehabilitation visit will take place within 10-14 days of the procedure, with encouragement to begin the home exercise program within 48-72 hours post-procedure. Additionally, all participants will be offered optional rehabilitative and/or complementary techniques available as standard of care such as aquatics, yoga, biofeedback, and pain psychology support, based on availability and as SOC.

The day of the treatment/injection will be considered study time point 0. Participants will return to clinic for follow up visits at 1 month (+/- 7 days), 3 months (+/- 14 days), 6 months (+/- 14 days) postinjection for PRP participants. Control participants will be given the option to received PRP treatment at the 3-month visit (more below). If participants opt for the injection, they will also come for a visit at 3 months (+/- 14 days) and 6 months (+/- 14 days) post-PRP injection. If they do not opt for the PRP injection, they will come 6-month (+/- 14 days) post-saline injection. At each follow-up visit, participants will undergo a standard physical examination by the provider who did not do the procedure (i.e. the AI or PI within the pain clinic) and the participant will assess current pain and functional level using the Numeric Pain Rating Scale (NRS-Pain) and the Defense Veteran Pain Rating Scale (DVPRS) Supplemental Questions.

Participants will also complete the Oswestry Disability Index (ODI), Global Rate of Change (GROC), PROMIS Pain Interference, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to participate in Social Roles and Activities, and the Work Productivity and Activity Impairment Questionnaire for Low Back Pain (WPAI:LBP). At each follow up visit, participants will be evaluated for adverse events and any additional treatment, therapy, and concomitant medications will be documented.

Study Blinding:

Participants will be blinded to assigned treatment arm (i.e. saline vs. PRP) until 3 months post-injection. Blinding will be revealed to participants at the end of their 3 month post-injection follow up visit after they complete all required follow up questionnaires. At this time, participants assigned to the control (saline injection) arm will be offered the option to receive PRP injections. Control participants who elect to receive PRP injections will remain in the study and will continue follow up with the research team until 6-months post PRP injection. Control participants that do not opt to receive PRP-injection at the 3- months post-saline injection, will remain in the study until 6 months post saline-injection.

Control participants who are not interested in receiving PRP injections and that would like to be treated with additional medical management (i.e. radiofrequency ablation) will resume normal care with their attending physician who will guide additional treatment options. Participants electing not to receive PRP will still be evaluated at 6-months post-injection visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-75 (inclusive)
* DEERS eligible
* Able to understand, read and speak English
* Willing and able to provide written informed consent
* Predominant area of pain is axial low back pain
* Chronic low back pain lasting more than 3 months
* Average daily numerical pain rating of at least 4 out of 10
* Single positive diagnostic medial branch block (MBB) of greater than or equal to 50% reduction in symptoms after local anesthetic injection

Exclusion Criteria:

* Prior spinal intervention such as epidural steroid injection or sacroiliac joint injection for current symptoms
* Prior radiofrequency denervation for facet mediated pain
* History of lumbar fusion
* Allergic to local anesthetic such as lidocaine and ropivacaine
* On opioid medication greater than or equal to 50 MME
* Recent (within past 3 months) systematic or localized infection
* Spinal pathology such as symptomatic radiculopathy or spinal stenosis within the past 3 months
* Medical or psychological condition that would preclude safe participation in study procedures (e.g. uncontrolled coagulopathy, diabetes, uncontrolled immunosuppression, inflammatory arthritis, active malignancy, uncontrolled depression or anxiety, etc.)
* Service member currently going through medical evaluation board
* Scheduled to move, deploy, separate or retire within 6 months
* Unable or unwilling to comply with study requirements
* Currently pregnant or had a recent delivery (within past 3 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 3 months
  Assesses average daily pain on a scale from 0-10

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | 6 months
  Assesses average daily pain on a scale from 0-10
Defense Veteran Pain Rating Scale+ Supplemental Questions (DVPRS) | 3 and 6 months
  Assesses for cognitive behavioral impacts of pain scale from 0-10
Oswestry Disability Index (ODI) | 3 and 6 months
  Assesses low back pain functional status changes scale from 0-10
Global Rate of Change (GROC) | 3 and 6 months
  Assesses change of the condition since the procedure
Patient Reported Outcomes Measurement Information System 29 and derived Pain Impact Scale(PROMIS-29) | 3 and 6 months
  Assesses pain impact changes scale from 0-10
Work Productivity and Activity Impairment Questionnaire for Low Back Pain (WPAI:LB) | 3 and 6 months
  Assesses work and activity impairment due to pain scale from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Min Ho Chang, MD, Principal Investigator — Womack Army Medical Center
Locations (1):
- Womack Army Medical Center, Fort Liberty, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Result] Dieleman JL, Baral R, Birger M, Bui AL, Bulchis A, Chapin A, Hamavid H, Horst C, Johnson EK, Joseph J, Lavado R, Lomsadze L, Reynolds A, Squires E, Campbell M, DeCenso B, Dicker D, Flaxman AD, Gabert R, Highfill T, Naghavi M, Nightingale N, Templin T, Tobias MI, Vos T, Murray CJ. US Spending on Personal Health Care and Public Health, 1996-2013. JAMA. 2016 Dec 27;316(24):2627-2646. doi: 10.1001/jama.2016.16885. PMID 28027366
- [Result] Jensen MC, Brant-Zawadzki MN, Obuchowski N, Modic MT, Malkasian D, Ross JS. Magnetic resonance imaging of the lumbar spine in people without back pain. N Engl J Med. 1994 Jul 14;331(2):69-73. doi: 10.1056/NEJM199407143310201. PMID 8208267
- [Result] Schwarzer AC, Wang SC, Bogduk N, McNaught PJ, Laurent R. Prevalence and clinical features of lumbar zygapophysial joint pain: a study in an Australian population with chronic low back pain. Ann Rheum Dis. 1995 Feb;54(2):100-6. doi: 10.1136/ard.54.2.100. PMID 7702395
- [Result] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Result] Manchikanti L, Kaye AD, Boswell MV, Bakshi S, Gharibo CG, Grami V, Grider JS, Gupta S, Jha SS, Mann DP, Nampiaparampil DE, Sharma ML, Shroyer LN, Singh V, Soin A, Vallejo R, Wargo BW, Hirsch JA. A Systematic Review and Best Evidence Synthesis of the Effectiveness of Therapeutic Facet Joint Interventions in Managing Chronic Spinal Pain. Pain Physician. 2015 Jul-Aug;18(4):E535-82. PMID 26218948
- [Result] Vekaria R, Bhatt R, Ellard DR, Henschke N, Underwood M, Sandhu H. Intra-articular facet joint injections for low back pain: a systematic review. Eur Spine J. 2016 Apr;25(4):1266-81. doi: 10.1007/s00586-016-4455-y. Epub 2016 Feb 23. PMID 26906169
- [Result] Lakemeier S, Lind M, Schultz W, Fuchs-Winkelmann S, Timmesfeld N, Foelsch C, Peterlein CD. A comparison of intraarticular lumbar facet joint steroid injections and lumbar facet joint radiofrequency denervation in the treatment of low back pain: a randomized, controlled, double-blind trial. Anesth Analg. 2013 Jul;117(1):228-35. doi: 10.1213/ANE.0b013e3182910c4d. Epub 2013 Apr 30. PMID 23632051
- [Result] Wu J, Du Z, Lv Y, Zhang J, Xiong W, Wang R, Liu R, Zhang G, Liu Q. A New Technique for the Treatment of Lumbar Facet Joint Syndrome Using Intra-articular Injection with Autologous Platelet Rich Plasma. Pain Physician. 2016 Nov-Dec;19(8):617-625. PMID 27906940
- [Result] Wu J, Zhou J, Liu C, Zhang J, Xiong W, Lv Y, Liu R, Wang R, Du Z, Zhang G, Liu Q. A Prospective Study Comparing Platelet-Rich Plasma and Local Anesthetic (LA)/Corticosteroid in Intra-Articular Injection for the Treatment of Lumbar Facet Joint Syndrome. Pain Pract. 2017 Sep;17(7):914-924. doi: 10.1111/papr.12544. Epub 2017 Feb 22. PMID 27989008
- [Result] LaPrade RF, Geeslin AG, Murray IR, Musahl V, Zlotnicki JP, Petrigliano F, Mann BJ. Biologic Treatments for Sports Injuries II Think Tank-Current Concepts, Future Research, and Barriers to Advancement, Part 1: Biologics Overview, Ligament Injury, Tendinopathy. Am J Sports Med. 2016 Dec;44(12):3270-3283. doi: 10.1177/0363546516634674. Epub 2016 Mar 29. PMID 27159318
- [Result] Murray IR, Geeslin AG, Goudie EB, Petrigliano FA, LaPrade RF. Minimum Information for Studies Evaluating Biologics in Orthopaedics (MIBO): Platelet-Rich Plasma and Mesenchymal Stem Cells. J Bone Joint Surg Am. 2017 May 17;99(10):809-819. doi: 10.2106/JBJS.16.00793. PMID 28509821
- [Result] Zlotnicki JP, Geeslin AG, Murray IR, Petrigliano FA, LaPrade RF, Mann BJ, Musahl V. Biologic Treatments for Sports Injuries II Think Tank-Current Concepts, Future Research, and Barriers to Advancement, Part 3: Articular Cartilage. Orthop J Sports Med. 2016 Apr 15;4(4):2325967116642433. doi: 10.1177/2325967116642433. eCollection 2016 Apr. PMID 27123466
- [Result] Hauret KG, Pacha L, Taylor BJ, Jones BH. Surveillance of Disease and Nonbattle Injuries During US Army Operations in Afghanistan and Iraq. US Army Med Dep J. 2016 Apr-Sep;(2-16):15-23. PMID 27215861
- [Result] Hauret KG, Jones BH, Bullock SH, Canham-Chervak M, Canada S. Musculoskeletal injuries description of an under-recognized injury problem among military personnel. Am J Prev Med. 2010 Jan;38(1 Suppl):S61-70. doi: 10.1016/j.amepre.2009.10.021. PMID 20117601

DOCUMENTS (1):
  • Informed Consent Form (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04822753/ICF_001.pdf